CLINICAL TRIAL: NCT06644950
Title: Efficacy and Safety of Administration of Different Doses of 4% Articaine (1:100,000 Epinephrine) Using the Lower Dental Nerve Block Technique for Lower Third Molar Extraction. a Triple-blind Randomized Clinical Trial.
Brief Title: Efficacy and Safety of Administration of Different Doses of 4% Articaine.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Adrià Jorba García, Prof. dr (DDS, MS,PhD), University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28/2022
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2022-10

CONDITIONS: Tooth Extraction Status Nos; Anesthesia, Local
Keywords: anesthesia; block nerve; wisdom tooth; wisdom tooth extraction

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two cartridges of anesthetic (Experimental): Two anesthetic cartridges of articaine 4% 1:100,000 will be administered with the direct technique for the inferior alveolar nerve block.
  Interventions: Other: Efficacy and safety of administering 1 or two cartridges of anesthesia
- Single cartridge of anesthetic (Active Comparator): In the control group, a single cartridge of anesthetic (1.8 mL of articaine 4% 1:100,000) will be injected and a second puncture will be simulated, contacting the syringe without needle, in the same area, counting up to 30 seconds.
  Interventions: Other: Efficacy and safety of administering 1 or two cartridges of anesthesia

INTERVENTIONS:
Other: Efficacy and safety of administering 1 or two cartridges of anesthesia — The investigator will administer the first anesthesia for NDI block with a cartridge of 4% articaine anesthetic at 1:100,000 . At the end, an envelope containing the assignment to the experimental or control group will be opened.
  In the control group, only the first anesthetic (1.8 mL of articaine 4% 1:100,000) will be injected and a second puncture will be simulated, contacting the syringe without the needle, in the same area, counting up to 30 seconds.
  In the experimental group two anesthetic cartridges of articaine 4% 1:100,000 will be administered with the direct technique for the inferior alveolar nerve block.

SUMMARY:
The goal of this triple-blind randomized clinical trial is to compare the efficacy and safety of administering one cartridge (1.8 mL) versus two cartridges of articaine 4% with epinephrine 1:100,000 for lower third molar extraction using the inferior alveolar nerve block technique.

The main questions it aims to answer are:

* The injection of 3.6 ml of 4% articaine 1:100,000 has a higher anesthetic efficacy than a single injection of 1.8 ml of the same anesthetic.
* The injection of 3.6 ml of 4% articaine 1:100,000 has a higher rate of adverse effects than a single injection of 1.8 ml of the same anesthetic.
* The injection of 3.6 ml of 4% articaine 1:100,000 has a greater alteration of heart rate, oxygen saturation and systolic and diastolic blood pressure than a single injection of 1.8 ml of the same anesthetic.

The investigator (XA) will perform the anesthetic technique.

* The investigator will administer a first anesthesia for NDI block with a cartridge of 4% articaine anesthetic at 1:100,000 . At the end, an envelope containing the assignment to the experimental or control group will be opened.

  * In the control group, a single cartridge of anesthetic (1.8 mL of articaine 4% 1:100,000) will be injected and a second puncture will be simulated, contacting the syringe without the needle, in the same area, counting up to 30 seconds.
  * In the experimental group two anesthetic cartridges of articaine 4% 1:100,000 will be administered with the direct technique for the inferior alveolar nerve block.
* After checking Vincent's sign, the vestibular (buccal nerve) infiltration will be performed in both groups with half a cartridge (0.9 ml) of the same anesthetic solution.
* The latency of the anesthetic effect will be measured using a pulpometer.
* Subsequently, a student of the Master's Degree in Oral Surgery of the University of Barcelona will perform the surgical intervention. The surgeons in charge of performing the extraction will not know to which group each patient belongs.
* The collection of the variables and the postoperative controls will be carried out by the researcher who has not performed the anesthetic technique and who will not know the study group to which the patient belongs.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥18 years) requiring surgical extraction of a lower wisdom tooth (whether erupted, semi-erupted or included).
* Patients without relevant systemic pathology (equal or lower than ASA II).
* Sufficient intellectual capacity to understand the study, the informed consent and to adequately complete the questionnaires.

Exclusion Criteria:

* Pregnant patients.
* Patients with hypersensitivity to articaine or adrenaline.
* Patients with uncontrolled systemic diseases.
* Drugs or systemic diseases (ASA III or higher) and that contraindicate a surgical intervention or the use of anesthetics and/or vasoconstrictors.
* Patients with relative or absolute contraindication of conventional analgesic or anti-inflammatory regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of administering one or two cartridges of articaine 4% with epinephrine 1:100,000 using the direct approach of the lower dental nerve block | 1 hour
  Determined by:
  * Achieving Vincent's sign within 6 minutes after injection.
  * Reporting a negative response to the pulpometer within 6 minutes after injection.
  * Absence of need for reanesthesia during the surgical procedure.

SECONDARY OUTCOMES:
To compare the safety of both techniques | 7 days
  Determined by the appearance or absence of adverse effects, such as : Disorientation, dizziness, blurred vision, nausea, vomiting, tremors, convulsions, vasovagal syncope, paresthesia or trismus.
Determine the hemodynamic changes that occur during surgery. | 1 to 2 hours
  Determined by the changes between the preoperative measurements and the postoperatives.

OTHER OUTCOMES:
Post-operative pain | 7 days
  Using a visual analog pain score from 0 to 10 centimeters at 2, 6, and 12 hours postoperatively and then daily until the seventh day after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Odontológic de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duarte-Rodrigues L, Miranda EFP, Souza TO, de Paiva HN, Falci SGM, Galvao EL. Third molar removal and its impact on quality of life: systematic review and meta-analysis. Qual Life Res. 2018 Oct;27(10):2477-2489. doi: 10.1007/s11136-018-1889-1. Epub 2018 May 24. PMID 29797177
- [Background] Ku JK, Kim JY, Jun MK, Jeong YK, Huh JK. Influence of General and Local Anesthesia on Postoperative Pain after Impacted Third Molar Surgery. J Clin Med. 2021 Jun 17;10(12):2674. doi: 10.3390/jcm10122674. PMID 34204470
- [Background] Sainz de Baranda B, Silvestre FJ, Silvestre-Rangil J. Relationship Between Surgical Difficulty of Third Molar Extraction Under Local Anesthesia and the Postoperative Evolution of Clinical and Blood Parameters. J Oral Maxillofac Surg. 2019 Jul;77(7):1337-1345. doi: 10.1016/j.joms.2019.02.020. Epub 2019 Feb 20. PMID 30878593
- [Background] Olmedo-Gaya MV, Manzano-Moreno FJ, Munoz-Lopez JL, Vallecillo-Capilla MF, Reyes-Botella C. Double-blind, randomized controlled clinical trial on analgesic efficacy of local anesthetics articaine and bupivacaine after impacted third molar extraction. Clin Oral Investig. 2018 Dec;22(9):2981-2988. doi: 10.1007/s00784-018-2386-1. Epub 2018 Feb 15. PMID 29450738
- [Background] Camps-Font O, Figueiredo R, Sanchez-Torres A, Cle-Ovejero A, Coulthard P, Gay-Escoda C, Valmaseda-Castellon E. Which is the most suitable local anaesthetic when inferior nerve blocks are used for impacted mandibular third molar extraction? A network meta-analysis. Int J Oral Maxillofac Surg. 2020 Nov;49(11):1497-1507. doi: 10.1016/j.ijom.2020.04.016. Epub 2020 May 27. PMID 32473767
- [Background] Santos-Sanz L, Toledano-Serrabona J, Gay-Escoda C. Safety and efficacy of 4% articaine in mandibular third-molar extraction: A systematic review and meta-analysis of randomized clinical trials. J Am Dent Assoc. 2020 Dec;151(12):912-923.e10. doi: 10.1016/j.adaj.2020.08.016. PMID 33228884
- [Background] Madan N, Shashidhara Kamath K, Gopinath AL, Yashvanth A, Vaibhav N, Praveen G. A Randomized Controlled Study Comparing Efficacy of Classical and Gow-Gates Technique for Providing Anesthesia During Surgical Removal of Impacted Mandibular Third Molar: A Split Mouth Design. J Maxillofac Oral Surg. 2017 Jun;16(2):186-191. doi: 10.1007/s12663-016-0960-0. Epub 2016 Sep 15. PMID 28439159
- [Background] Montserrat-Bosch M, Figueiredo R, Nogueira-Magalhaes P, Arnabat-Dominguez J, Valmaseda-Castellon E, Gay-Escoda C. Efficacy and complications associated with a modified inferior alveolar nerve block technique. A randomized, triple-blind clinical trial. Med Oral Patol Oral Cir Bucal. 2014 Jul 1;19(4):e391-7. doi: 10.4317/medoral.19554. PMID 24608204
- [Background] Figueiredo R, Sofos S, Soriano-Pons E, Camps-Font O, Sanmarti-Garcia G, Gay-Escoda C, Valmaseda-Castellon E. Is it possible to extract lower third molars with infiltration anaesthesia techniques using articaine? A double-blind randomized clinical trial. Acta Odontol Scand. 2021 Jan;79(1):1-8. doi: 10.1080/00016357.2020.1760348. Epub 2020 May 13. PMID 32401086
- [Background] Kim C, Hwang KG, Park CJ. Local anesthesia for mandibular third molar extraction. J Dent Anesth Pain Med. 2018 Oct;18(5):287-294. doi: 10.17245/jdapm.2018.18.5.287. Epub 2018 Oct 31. PMID 30402548
- [Background] Madan GA, Madan SG, Madan AD. Failure of inferior alveolar nerve block: exploring the alternatives. J Am Dent Assoc. 2002 Jul;133(7):843-6. doi: 10.14219/jada.archive.2002.0298. PMID 12148677
- [Background] Yang F, Gao Y, Zhang L, Zheng B, Wang L, Sun H, Huang D. Local anaesthesia for surgical extraction of mandibular third molars: a systematic review and network meta-analysis. Clin Oral Investig. 2020 Nov;24(11):3781-3800. doi: 10.1007/s00784-020-03490-3. Epub 2020 Aug 24. PMID 32833132
- [Background] Sawang K, Chaiyasamut T, Kiattavornchareon S, Pairuchvej V, Bhattarai BP, Wongsirichat N. Double versus single cartridge of 4% articaine infiltration into the retro-molar area for lower third molar surgery. J Dent Anesth Pain Med. 2017 Jun;17(2):121-127. doi: 10.17245/jdapm.2017.17.2.121. Epub 2017 Jun 29. PMID 28879339
- [Background] Renton T, Janjua H, Gallagher JE, Dalgleish M, Yilmaz Z. UK dentists' experience of iatrogenic trigeminal nerve injuries in relation to routine dental procedures: why, when and how often? Br Dent J. 2013 Jun;214(12):633-42. doi: 10.1038/sj.bdj.2013.583. PMID 23787854
- [Background] Hillerup S, Jensen R. Nerve injury caused by mandibular block analgesia. Int J Oral Maxillofac Surg. 2006 May;35(5):437-43. doi: 10.1016/j.ijom.2005.10.004. Epub 2005 Dec 15. PMID 16343853
- [Background] Haas DA, Lennon D. A 21 year retrospective study of reports of paresthesia following local anesthetic administration. J Can Dent Assoc. 1995 Apr;61(4):319-20, 323-6, 329-30. PMID 7736335
- [Background] Garisto GA, Gaffen AS, Lawrence HP, Tenenbaum HC, Haas DA. Occurrence of paresthesia after dental local anesthetic administration in the United States. J Am Dent Assoc. 2010 Jul;141(7):836-44. doi: 10.14219/jada.archive.2010.0281. PMID 20592403
- [Background] Gaffen AS, Haas DA. Retrospective review of voluntary reports of nonsurgical paresthesia in dentistry. J Can Dent Assoc. 2009 Oct;75(8):579. PMID 19840499
- [Background] Sancho-Puchades M, Vilchez-Perez MA, Valmaseda-Castellon E, Paredes-Garcia J, Berini-Aytes L, Gay-Escoda C. Bupivacaine 0.5% versus articaine 4% for the removal of lower third molars. A crossover randomized controlled trial. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e462-8. doi: 10.4317/medoral.17628. PMID 22143739
- [Background] Abazarpoor R, Parirokh M, Nakhaee N, Abbott PV. A Comparison of Different Volumes of Articaine for Inferior Alveolar Nerve Block for Molar Teeth with Symptomatic Irreversible Pulpitis. J Endod. 2015 Sep;41(9):1408-11. doi: 10.1016/j.joen.2015.05.015. Epub 2015 Jul 3. PMID 26149210
- [Background] Fowler S, Reader A, Beck M. Incidence of missed inferior alveolar nerve blocks in vital asymptomatic subjects and in patients with symptomatic irreversible pulpitis. J Endod. 2015 May;41(5):637-9. doi: 10.1016/j.joen.2015.01.029. Epub 2015 Mar 11. PMID 25770038
- [Background] Malamed SF. Is the mandibular nerve block passe? J Am Dent Assoc. 2011 Sep;142 Suppl 3:3S-7S. doi: 10.14219/jada.archive.2011.0340. PMID 21881055
- [Background] Alvira-Gonzalez J, Figueiredo R, Valmaseda-Castellon E, Quesada-Gomez C, Gay-Escoda C. Predictive factors of difficulty in lower third molar extraction: A prospective cohort study. Med Oral Patol Oral Cir Bucal. 2017 Jan 1;22(1):e108-e114. doi: 10.4317/medoral.21348. PMID 27918736
- [Background] Garcia Garcia A, Gude Sampedro F, Gandara Rey J, Gallas Torreira M. Trismus and pain after removal of impacted lower third molars. J Oral Maxillofac Surg. 1997 Nov;55(11):1223-6. doi: 10.1016/s0278-2391(97)90172-5. PMID 9371111
- [Background] Rood JP, Shehab BA. The radiological prediction of inferior alveolar nerve injury during third molar surgery. Br J Oral Maxillofac Surg. 1990 Feb;28(1):20-5. doi: 10.1016/0266-4356(90)90005-6. PMID 2322523